CLINICAL TRIAL: NCT01625000
Title: A Double-Blind, Placebo-Controlled Study of MP-214 in Patients With Schizophrenia
Brief Title: Safety and Efficacy of MP-214 in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A002-A4
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Results first posted 2021-04-12 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Antipsychotic Agents; Acute Schizophrenia; Mental Disorder; Psychotropic Drugs; Dopamine Agents; Risperidone; Central Nervous System Agents
MeSH Terms: conditions — Schizophrenia; Mental Disorders | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- MP-214 3mg (Experimental)
  Interventions: Drug: MP-214 3mg
- MP-214 6mg (Experimental)
  Interventions: Drug: MP-214 6mg
- MP-214 9mg (Experimental)
  Interventions: Drug: MP-214 9mg
- Risperidone 4mg (Active Comparator)
  Interventions: Drug: Risperidone 4mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MP-214 3mg — Patients who meet eligibility criteria will be administered a once daily oral 3mg of MP-214 for six weeks.
  Arms: MP-214 3mg
Drug: MP-214 6mg — Patients who meet eligibility criteria will be administered a once daily oral 6mg of MP-214 for six weeks.
  Arms: MP-214 6mg
Drug: MP-214 9mg — Patients who meet eligibility criteria will be administered a once daily oral 9mg of MP-214 for six weeks.
  Arms: MP-214 9mg
Drug: Risperidone 4mg — Patients who meet eligibility criteria will be administered a once daily oral 4mg of risperidone for six weeks.
  Arms: Risperidone 4mg
Drug: Placebo — Patients who meet eligibility criteria will be administered a once daily oral dose of placebo for six weeks.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy, safety, and tolerability of MP-214 relative to placebo in patients with acute exacerbation of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient before the initiation of any study-specific procedures
* Patients diagnosed with schizophrenia according to the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for schizophrenia
* Patients with normal physical examination, laboratory, vital signs, and/or electrocardiogram (ECG)

Exclusion Criteria:

* Patients with a DSM-IV-TR diagnosis of schizoaffective disorder, schizophreniform disorder, other psychotic disorders other than schizophrenia, or bipolar I or II disorder

The information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 512 (Actual)
Dates: Start 2012-05; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Sapporo, Hokkaido, Japan
- Seoul, South Korea
- Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four subjects withdrew from the study before the start of the study medication after being assigned to the treatment.
Period: Overall Study
Arm/Group | MP-214 3mg | MP-214 6mg | MP-214 9mg | Risperidone 4mg | Placebo
Started | 126 | 133 | 67 | 56 | 126
Completed | 74 | 81 | 34 | 37 | 71
Not Completed | 52 | 52 | 33 | 19 | 55
Not completed — Physician Decision | 15 | 7 | 7 | 2 | 15
Not completed — Protocol Violation | 3 | 10 | 4 | 1 | 2
Not completed — Withdrawal by Subject | 19 | 16 | 11 | 9 | 17
Not completed — Adverse Event (including Death) | 15 | 19 | 11 | 7 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MP-214 3mg | MP-214 6mg | MP-214 9mg | Risperidone 4mg | Placebo | Total
Number analyzed (Participants) | 126 | 133 | 67 | 56 | 126 | 508
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (10.6) | 40.2 (11.4) | 43.0 (9.7) | 39.5 (10.2) | 40.1 (11.1) | 40.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 34 | 25 | 66 | 245
  Male | 66 | 73 | 33 | 31 | 60 | 263

OUTCOME MEASURES:

1. Primary Outcome: Change in the Positive and Negative Syndrome Scale (PANSS) Total Score at Week 6
Description: PANSS score is a 30-item rating scale to assess both the positive and negative symptom syndromes of patients with schizophrenia. Each item is scored on a 7-point scale, from 1 (absent) to 7 (extreme). The PANSS total score of the 30 PANSS items ranges from 30 to 210. High scores indicate greater severity of symptoms.
Time Frame: Baseline and Week 6
Population: For OC (Observed Case) analysis, the Missing Values were Not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | MP-214 3mg | MP-214 6mg | MP-214 9mg | Risperidone 4mg | Placebo
Number analyzed (Participants) | 78 | 80 | 36 | 36 | 71
units on a scale | -10.4 (2.0) | -13.8 (2.0) | -14.0 (2.9) | -20.2 (3.0) | -9.5 (2.1)

2. Secondary Outcome: Change in the Clinical Global Impression-Severity (CGI-S) Score at Week 6
Description: CGI-S is a 7-point scale to assess the global severity of the participant's illness. CGI-S scores range from 1 (normal, not ill at all) to 7 (extremely ill).
Time Frame: Baseline and Week 6
Population: For OC (Observed Case) analysis, the Missing Values were Not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | MP-214 3mg | MP-214 6mg | MP-214 9mg | Risperidone 4mg | Placebo
Number analyzed (Participants) | 78 | 80 | 36 | 36 | 71
units on a scale | -0.7 (0.1) | -0.8 (0.1) | -0.7 (0.2) | -1.2 (0.2) | -0.6 (0.1)

ADVERSE EVENTS:
Arm/Group | MP-214 3mg | MP-214 6mg | MP-214 9mg | Risperidone 4mg | Placebo
Serious Adverse Events (participants affected / at risk) | 12/126 | 16/133 | 4/67 | 2/56 | 14/126
Other Adverse Events (participants affected / at risk) | 95/126 | 100/133 | 52/67 | 36/56 | 72/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MP-214 3mg (N=126) | MP-214 6mg (N=133) | MP-214 9mg (N=67) | Risperidone 4mg (N=56) | Placebo (N=126)
Sudden death (General disorders) | 0 | 1 | 0 | 0 | 0
Infection masked (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neuroleptic malignant syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 9 | 14 | 3 | 0 | 12
Suicidal behaviour (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MP-214 3mg (N=126) | MP-214 6mg (N=133) | MP-214 9mg (N=67) | Risperidone 4mg (N=56) | Placebo (N=126)
Constipation (Gastrointestinal disorders) | 21 | 20 | 12 | 5 | 15
Diarrhoea (Gastrointestinal disorders) | 6 | 8 | 4 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 4 | 4 | 2 | 3
Nausea (Gastrointestinal disorders) | 15 | 9 | 7 | 4 | 5
Vomiting (Gastrointestinal disorders) | 18 | 12 | 5 | 1 | 7
Nasopharyngitis (Infections and infestations) | 10 | 15 | 9 | 8 | 6
Contusion (Injury, poisoning and procedural complications) | 4 | 3 | 2 | 2 | 8
Blood creatine phosphokinase increased (Investigations) | 7 | 5 | 0 | 2 | 5
Liver function test abnormal (Investigations) | 1 | 1 | 5 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 6 | 7 | 2 | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 3 | 1
Akathisia (Nervous system disorders) | 28 | 19 | 2 | 9 | 10
Dizziness (Nervous system disorders) | 4 | 6 | 3 | 4 | 4
Extrapyramidal disorder (Nervous system disorders) | 11 | 19 | 11 | 6 | 12
Headache (Nervous system disorders) | 19 | 14 | 7 | 4 | 14
Somnolence (Nervous system disorders) | 3 | 2 | 5 | 1 | 3
Tremor (Nervous system disorders) | 7 | 13 | 1 | 0 | 4
Insomnia (Psychiatric disorders) | 12 | 16 | 5 | 2 | 9
Restlessness (Psychiatric disorders) | 3 | 5 | 4 | 3 | 5
Schizophrenia (Psychiatric disorders) | 16 | 15 | 13 | 7 | 23
Hypertension (Vascular disorders) | 0 | 5 | 6 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other